CLINICAL TRIAL: NCT01637428
Title: The Use of Intermittent Pneumatic Compression Device for Symptomatic Relief in Patients With Post Thrombotic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Galia Spectre, MD, Hadassah Medical Organization
Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 727209-HMO-CTIL
Record Dates: First submitted 2012-06-13; First posted 2012-07-11 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Post Thrombotic Syndrome
MeSH Terms: conditions — Postthrombotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ActiveCare+S.F.T 3rd generation — Intermittent Pneumatic Compression Device

SUMMARY:
The use of ActiveCare+S.F.T 3rd generation (an Intermittent Pneumatic Compression Device) will improve quality of life in patients suffering from Post Thrombotic Syndrome compared to compression stockings which is the current gold standard of care.

ELIGIBILITY:
Inclusion Criteria:

* patients who have developed post Thrombotic leg symptoms after a deep vein thrombosis event.

Exclusion Criteria:

* admitted patients
* Patients who suffer from peripheral artery disease.
* Patients with an acute deep vein thrombosis.
* s/p leg skin transplant
* Patients with an active leg infection
* Patients who aren't capable of operating the device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Quality of life (Veins-QOL) | 1 month

SECONDARY OUTCOMES:
Villalta Scale | 1 month
  The scale consists of five patient-rated venous symptoms (pain, cramps, heaviness, paresthesia, pruritus) and six clinician-rated physical signs (pretibial edema, skin induration, hyperpigmentation,pain during calf compression, venous ectasia, redness),which are each rated on a four-point scale (0 = none,1 = mild, 2 = moderate, 3 = severe). Points are summed to produce a total score (range: 0-33). Subjects are classified as having Post Thrombotic Syndrome if the score is 5 or more, or if a venous ulcer is present, in a leg with previous DVT.

CONTACTS AND LOCATIONS:
Overall Officials: Galia Spectre, MD, Principal Investigator — Hematology departement, Haddash medical Center, Jerusalem, Israel
Locations (1):
- Hadassah Ein Karem Medical Center, Jerusalem, Israel